CLINICAL TRIAL: NCT02442882
Title: The Acute Effect of Boxing on Balance, Neuropsychological, and Visual Functions
Status: Completed | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, David R Howell, Post-Doctoral Research Fellow, Boston Children's Hospital
Other Study IDs: IRB-P00018178
Record Dates: First submitted 2015-05-11; First posted 2015-05-13 (Estimated); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: Craniocerebral Trauma
Keywords: Brain Concussion; Balance; Locomotion; Mild Traumatic Brain Injury
MeSH Terms: conditions — Craniocerebral Trauma; Brain Concussion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Boxers: Individuals who participate in a boxing tournament will be tested on balance, neuropsychological, and visual functions before and after the tournament.

SUMMARY:
Prior research has investigated the effect of repetitive head trauma as it relates to physiological and psychological function. Boxing is one particular sport which predisposes athletes to a large amount of head impacts. We plan to assess the effects of a boxing tournament on balance, neuropsychological, and visual functions.

DETAILED DESCRIPTION:
This is a prospective, repeated measures cohort study, which is able to make within-subject (pre and post boxing tournament) comparisons on measures of physiologic and behavioral function.

We plan to enroll boxing athletes who are participating in a boxing tournament. Each individual will be assessed on the following tests: balance (dynamic and static balance), vestibular-ocular motor function, neuropsychological function, and symptoms. Additionally, each boxing match will be video recorded and the total number of head impacts they sustain will be documented.

* In order to prospectively assess how a boxing tournament affects balance, neuropsychological, and visual functions from pre-tournament assessments to post-tournament assessments (Specific Aim 1), we plan to test all athletes before competition at the Pan-American games begins (pre-test) and after they have been eliminated from the tournament (post-test).
* In order to measure the associations between the number of head blows sustained during a boxing tournament with balance, neuropsychological, visual, and symptom deficits, we will also use a video camera to record each match and count the total number of hits to the head.

ELIGIBILITY:
Inclusion Criteria:

1. Participation in boxing at a pre-specified tournament
2. Medically cleared to participate in the tournament, as determined by the attending medical staff

Exclusion Criteria:

1. Any pre-existing neurological disorder, including but not limited to stroke, intracranial hemorrhage, any movement disorder, and cerebral palsy.
2. Any currently active psychiatric condition, including specifically major depression, bipolar disorder or schizophrenia. A history of a psychiatric condition but no ongoing psychiatric episode (e.g. not currently undergoing treatment for a major depressive episode) would not be an exclusion.
3. Any unstable medical condition

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients will be recruited from those who are participating at a boxing tournament.
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2016-07; Primary Completion 2017-07-01 (Actual); Study Completion 2017-07-01 (Actual)

PRIMARY OUTCOMES:
Balance Control | 1 week
  Pre-tournament and post-tournament assessment of balance

SECONDARY OUTCOMES:
Neuropsychological function | 1 week
  Pre-tournament and post-tournament assessment of neuropsychological function
Visual function | 1 week
  Pre-tournament and post-tournament assessment of visual function

CONTACTS AND LOCATIONS:
Overall Officials: William P Meehan III, MD, Principal Investigator — Boston Children's Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Howell DR, Meehan WP 3rd, Loosemore MP, Cummiskey J, Grabner von Rosenberg JP, McDonagh D. Neurological tests improve after Olympic-style boxing bouts: a pretournament and post-tournament study in the 2016 Women's World Boxing Championships. Br J Sports Med. 2017 Sep;51(17):1279-1284. doi: 10.1136/bjsports-2016-097160. Epub 2017 May 13. PMID 28501805